CLINICAL TRIAL: NCT03763617
Title: Periosteal Inhibition Technique for Ridge Preservation A Prospective Study
Acronym: PI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinique Dentaire et d'implantologie Dr.Vinh Nguyen (Other)
Collaborators: Goethe University (Other)
Responsible Party: Principal Investigator, Vinh Giap Nguyen, DDS, Principal investigator, Clinique Dentaire et d'implantologie Dr.Vinh Nguyen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI2018
Record Dates: First submitted 2018-12-01; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Ridge Deficency
Keywords: Socket preservation

STUDY DESIGN:
Intervention Model Description: A d-ptfe membrane is placed between the buccal bone and periosteum of an extraction socket to prevent the precursors of the bone resorbing cells (osteoclasts) from adhering to the bone surface.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): A d-ptfe membrane will be placed between the buccal bone and periosteum of an extraction socket during a 4 months healing time before it is surgically removed.
  Interventions: Device: d-ptfe membrane
- Control group (No Intervention): The extraction socket will be left to heal naturally without a socket preservation intervention.

INTERVENTIONS:
Device: d-ptfe membrane — Socket preservation using d-ptfe membrane to inhibit the formation of osteoclasts
  Arms: Test group

SUMMARY:
The efficacy of the Periosteal Inhibition technique for socket preservation is studies against a control group in which the extraction sockets are allowed to heal without a socket preservation procedure.

DETAILED DESCRIPTION:
Socket preservation procedures have been shown to significantly reduce the loss of ridge dimension of an extraction socket. These procedures involve filling the empty socket with a bone graft material, which, serves as scaffold to limit horizontal and vertical ridge alterations. In order to contain the graft material, an occlusive barrier such as an autogenous soft tissue graft, resorbable or non-resorbable membrane, is often required. As yet, no one socket preservation technique has been proven superior to another, and none have proven totally effective in preserving ridge morphology. A net reduction of 1.5 mm in ridge width and 0.5 mm in ridge height is often observed after socket preservation procedures, which may necessitate additional hard or soft tissue augmentation to fully restore the ridge dimension.

In an animal histologic study in 2005, Araujo and Lindhe demonstrated that trauma and loss of periodontal ligament triggered an osteoclastic activity causing loss of bundle bone and modeling of the cortical bone plate. Osteoclasts are multi-nucleated cells that are responsible for bone resorption and are found on the outer layer of bone, beneath the periosteum. Osteoclasts are thought to be derived from pluripotent hematopoietic stem cells. When stimulated, these mononuclear precursors, the smallest of which is 9.5 microns in diameter, proliferate and attach to the bone surface to be resorbed, and only then fuse to form large mature multinucleated osteoclasts.

High-density polytetrafluoroethylene (d-ptfe) membranes have been used in socket preservation procedures as an occlusive barrier to contain the bone graft material.Polytetrafluoroethylene, a stable polymer and highly biocompatible, has a membrane porosity of less than 0.3 microns. It is impervious to bacteria and thus is recommended for a socket preservation technique, where a membrane is intentionally exposed.

In the present study, a high-density polytetrafluoroethylene (d-ptfe) membrane is placed between the periosteum and the buccal bone plate of an extraction socket where it will stay for a duration of 4 months, the time needed for the completion of bone forming within the socket. The goal of the non-resorbable d-ptfe membrane is to prevent the migration of precursor cells to the bone surface and thus their fusion to form osteoclast. The authors hypothesize that the passage of the precursor cells from the periosteum to the bone surface is inhibited by the small-diameter pores in the non-resorbable d-ptfe membrane. Osteolytic activity on the outer surface of the socket is thereby prevented as the precursor cells cannot form osteoclasts. The author coins the term "Periosteal Inhibition technique" for this socket preservation procedure.The study will compare dimension changes between extraction socket treated using the Periosteal Inhibition technique and those allowed to heal without a socket preservation procedure.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age
* Systemically healthy
* An extraction of one non-salvageable molar or premolar tooth is indicated. Adjacent teeth must be present to support the measuring template.
* Demonstrated ability to maintain goodoral hygiene
* Willingness and ability to commit to follow-up
* Able to understand study procedure and provide signed informed consent.

Exclusion Criteria:

* Extensive damaged buccal or lingual bone plate
* Extreme alveolar ridge atrophy
* Extensive vertical bone loss
* Active infection at the extraction site
* Uncontrolled periodontal disease.
* Recent febrile illness (within 6 months) that precludes or delays participation
* Severe renal or liver diseases
* History of radiotherapy of the head and neck region
* Chemotherapy for treatment of malignant tumors at the time of the study.
* Immuno-compromised patients
* Patients on IV bisphosphonates or on long term oral bisphosphonates for more than 3 years.
* Use of disallowed concomitant medications.
* Pregnancy or intending to conceive during the course of the Study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Ridge widths | 0 hour and 4 months
  Bucco-lingual ridge dimensions at the midline is measured at 3mm and 5mm apical to the gingival margin, at the time of extraction intra-op and 4 months post-extraction, using a acrylic template for repeatable measurements.
Change in Ridge widths on the buccal and lingual aspects | 0 hour and 4 months
  Buccal and lingual ridge dimension change at the midline is measured at 3mm and 5mm apical to the gingival margin, at the time of extraction and 4 months post-extraction, using a acrylic template for repeatable measurements.
Change in Ridge heights | 0 hour and 4 months
  Change in Ridge bone heights at messiah and distal interproximal, mid-buccal and mid-lingual aspects.

SECONDARY OUTCOMES:
Bone plate thickness | 0 hour
  Marginal buccal and lingual bone plate thickness
Keratinized mucosa | 0 hour and 4 months
  Width of keratinized mucosa over the ridge

OTHER OUTCOMES:
Complications | 1 month, 2 months, 3 months and 4 months
  To assess complication rate of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Vinh Giap Nguyen, DDS, MSc, Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Walker CJ, Prihoda TJ, Mealey BL, Lasho DJ, Noujeim M, Huynh-Ba G. Evaluation of Healing at Molar Extraction Sites With and Without Ridge Preservation: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):241-249. doi: 10.1902/jop.2016.160445. Epub 2016 Oct 27. PMID 27788625
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] MacBeth N, Trullenque-Eriksson A, Donos N, Mardas N. Hard and soft tissue changes following alveolar ridge preservation: a systematic review. Clin Oral Implants Res. 2017 Aug;28(8):982-1004. doi: 10.1111/clr.12911. Epub 2016 Jul 26. PMID 27458031
- [Background] Iocca O, Farcomeni A, Pardinas Lopez S, Talib HS. Alveolar ridge preservation after tooth extraction: a Bayesian Network meta-analysis of grafting materials efficacy on prevention of bone height and width reduction. J Clin Periodontol. 2017 Jan;44(1):104-114. doi: 10.1111/jcpe.12633. Epub 2016 Dec 5. PMID 27712001
- [Background] Willenbacher M, Al-Nawas B, Berres M, Kammerer PW, Schiegnitz E. The Effects of Alveolar Ridge Preservation: A Meta-Analysis. Clin Implant Dent Relat Res. 2016 Dec;18(6):1248-1268. doi: 10.1111/cid.12364. Epub 2015 Jul 1. PMID 26132885
- [Background] Hakeda Y, Kumegawa M. [Osteoclasts in bone metabolism]. Kaibogaku Zasshi. 1991 Aug;66(4):215-25. Japanese. PMID 1759556
- [Background] Hagenaars CE, van der Kraan AA, Kawilarang-de Haas EW, Visser JW, Nijweide PJ. Osteoclast formation from cloned pluripotent hemopoietic stem cells. Bone Miner. 1989 May;6(2):179-89. doi: 10.1016/0169-6009(89)90049-4. PMID 2788471
- [Background] Buckwalter JA, Glimcher MJ, Cooper RR, Recker R. Bone biology. I: Structure, blood supply, cells, matrix, and mineralization. Instr Course Lect. 1996;45:371-86. No abstract available. PMID 8727757
- [Background] Wagner JE, Collins D, Fuller S, Schain LR, Berson AE, Almici C, Hall MA, Chen KE, Okarma TB, Lebkowski JS. Isolation of small, primitive human hematopoietic stem cells: distribution of cell surface cytokine receptors and growth in SCID-Hu mice. Blood. 1995 Jul 15;86(2):512-23. PMID 7541665
- [Background] Baron R, Neff L, Tran Van P, Nefussi JR, Vignery A. Kinetic and cytochemical identification of osteoclast precursors and their differentiation into multinucleated osteoclasts. Am J Pathol. 1986 Feb;122(2):363-78. PMID 3946557
- [Background] Hoffmann O, Bartee BK, Beaumont C, Kasaj A, Deli G, Zafiropoulos GG. Alveolar bone preservation in extraction sockets using non-resorbable dPTFE membranes: a retrospective non-randomized study. J Periodontol. 2008 Aug;79(8):1355-69. doi: 10.1902/jop.2008.070502. PMID 18672984
- [Background] Laurito D, Cugnetto R, Lollobrigida M, Guerra F, Vestri A, Gianno F, Bosco S, Lamazza L, De Biase A. Socket Preservation with d-PTFE Membrane: Histologic Analysis of the Newly Formed Matrix at Membrane Removal. Int J Periodontics Restorative Dent. 2016 Nov/Dec;36(6):877-883. doi: 10.11607/prd.2114. PMID 27740650
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Camargo PM, Lekovic V, Carnio J, Kenney EB. Alveolar bone preservation following tooth extraction: a perspective of clinical trials utilizing osseous grafting and guided bone regeneration. Oral Maxillofac Surg Clin North Am. 2004 Feb;16(1):9-18, v. doi: 10.1016/j.coms.2003.10.004. PMID 18088709
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Serino G, Biancu S, Iezzi G, Piattelli A. Ridge preservation following tooth extraction using a polylactide and polyglycolide sponge as space filler: a clinical and histological study in humans. Clin Oral Implants Res. 2003 Oct;14(5):651-8. doi: 10.1034/j.1600-0501.2003.00970.x. PMID 12969370
- [Background] Guarnieri R, Aldini NN, Pecora G, Fini M, Giardino R. Medial-grade calcium sulfate hemihydrate (surgiplaster) in healing of a human extraction socket--histologic observation at 3 months: a case report. Int J Oral Maxillofac Implants. 2005 Jul-Aug;20(4):636-41. PMID 16161750
- [Background] Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets. Part 1: histomorphometric evaluations at 9 months. J Periodontol. 2000 Jun;71(6):1015-23. doi: 10.1902/jop.2000.71.6.1015. PMID 10914806
- [Background] Nappi JF, Lehman JA Jr. The effects of Surgicel on bone formation. Cleft Palate J. 1980 Oct;17(4):291-6. PMID 6934043
- [Background] Armstrong JK, Han B, Kuwahara K, Yang Z, Magyar CE, Dry SM, Atti E, Tetradis S, Fisher TC. The effect of three hemostatic agents on early bone healing in an animal model. BMC Surg. 2010 Dec 17;10:37. doi: 10.1186/1471-2482-10-37. PMID 21167039
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Sanz M, Cecchinato D, Ferrus J, Pjetursson EB, Lang NP, Lindhe J. A prospective, randomized-controlled clinical trial to evaluate bone preservation using implants with different geometry placed into extraction sockets in the maxilla. Clin Oral Implants Res. 2010 Jan;21(1):13-21. doi: 10.1111/j.1600-0501.2009.01824.x. Epub 2009 Nov 18. PMID 19922492
- [Background] Sanz M, Lindhe J, Alcaraz J, Sanz-Sanchez I, Cecchinato D. The effect of placing a bone replacement graft in the gap at immediately placed implants: a randomized clinical trial. Clin Oral Implants Res. 2017 Aug;28(8):902-910. doi: 10.1111/clr.12896. Epub 2016 Jun 7. PMID 27273298
- [Background] Chappuis V, Engel O, Shahim K, Reyes M, Katsaros C, Buser D. Soft Tissue Alterations in Esthetic Postextraction Sites: A 3-Dimensional Analysis. J Dent Res. 2015 Sep;94(9 Suppl):187S-93S. doi: 10.1177/0022034515592869. Epub 2015 Jun 30. PMID 26130259
- [Background] Chappuis V, Engel O, Reyes M, Shahim K, Nolte LP, Buser D. Ridge alterations post-extraction in the esthetic zone: a 3D analysis with CBCT. J Dent Res. 2013 Dec;92(12 Suppl):195S-201S. doi: 10.1177/0022034513506713. Epub 2013 Oct 24. PMID 24158340